CLINICAL TRIAL: NCT01202656
Title: G-CSF(Granulocyte Colony Stimulating Factor) and Embryo Implantation and Pregnancy Following IVF (in Vitro Fertilization)
Brief Title: Effect of Colony Stimulating Factor on Implantation and Pregnancy Rates Following IVF (in Vitro Fertilization)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Center for Human Reproduction (Other)
Collaborators: Foundation for Reproductive Medicine (Other)
Responsible Party: Principal Investigator, David H. Barad, Director of Clinical Research, Center for Human Reproduction
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09012010-02
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Results first posted 2014-12-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Infertility, Female
Keywords: Fertility Agents, Female; In vitro fertilization
MeSH Terms: conditions — Infertility, Female | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G-CSF then Saline (Experimental): G-CSF (Granulocyte colony stimulating factor)
  Interventions: Drug: G-CSF; Drug: Saline
- Saline then G-CSF (Placebo Comparator): Normal Saline
  Interventions: Drug: G-CSF; Drug: Saline

INTERVENTIONS:
Drug: G-CSF — One infusion of G-CSF 300 units administered by intrauterine infusion
  Other Names: Neupogen (Filgrastim)
Drug: Saline — intrauterine saline infusion 1 cc
  Other Names: Normal Saline; 0.91% w/v of NaCl, about 300 mOsm/L

SUMMARY:
This a trial designed to test whether granulocyte colony stimulating factor (G-CSF, Neupogen) can increase the rate of embryo implantation following IVF and embryo transfer. Preliminary data at the Center for Human Reproduction(CHR) and elsewhere suggest that intrauterine infusion of G-CSF can improve endometrial development and can increase implantation rates of embryos.

DETAILED DESCRIPTION:
Objective: To investigate the effect of treatment with CSF on pregnancy rates in routine in vitro fertilization (IVF).

Design: Double blinded crossover randomized controlled clinical trial

Setting: Academically affiliated private infertility centers

Subjects: Normal female IVF patients 18-38 years old, and above age 38 years, who are willing to be randomized to treatment.

Interventions: Subjects receive transvaginally, utilizing an insemination catheter, a slow uterine lavage with G-CSF (Neupogen), 300ug (in 1 ml); controls receive saline. Patients who do not conceive will, after one month washout time, continue treatment in the opposite study arm.

Main Outcome Measures: Implantation rate(IR) and pregnancy rates.

Second Outcome Measures: Live birth rates and miscarriage rates.

Statistical and Power considerations: Analysis will be by regression with IR as dependent and treatment as independent. Results will be adjusted by age and indices of ovarian reserve, such as antiMulerian Hormone (AMH). Presuming an implantation rate of 10% and anticipating a 10% increase to 20% with treatment, 120 women, producing about 200 embryos in each study arm, will have to be recruited for 80% power and alpha of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Women already enrolled in an IVF cycle at one of the participating institutions

Exclusion Criteria:

* Sickle Cell disease
* Renal insufficiency
* Upper respiratory infection or Pneumonia
* Chronic Neutropenia
* Known Past or present malignancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Barad, MD, MS, Principal Investigator — Center for Human Reproduction; Norbert Gleicher, MD, Study Chair — Center for Human Reproduction
Locations (1):
- Center for Human Reproduction, New York, New York, United States

REFERENCES:
- [Result] Barad DH, Yu Y, Kushnir VA, Shohat-Tal A, Lazzaroni E, Lee HJ, Gleicher N. A randomized clinical trial of endometrial perfusion with granulocyte colony-stimulating factor in in vitro fertilization cycles: impact on endometrial thickness and clinical pregnancy rates. Fertil Steril. 2014 Mar;101(3):710-5. doi: 10.1016/j.fertnstert.2013.12.016. Epub 2014 Jan 11. PMID 24424357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients presenting for embryos transfer between October 3, 2010, and January 1, 2013, were offered participation in the trial. A total of 419 eligible patients were offered participation: Only 129 patients consented to participate in this study,(12 addtional patient participated in the thin endometrium study) and 278 declined
Pre-assignment Details: The principal reasons for refusal to participate were ''lack of interest'' and technical difficulties in presenting in timely fashion for the treatment to the center. Women with renal disease, sickle cell disease, or a history of malignancy were considered ineligible. No consenting patient was excluded from participation for medical reasons.
Groups:
- G-CSF Then Saline: G-CSF (Granulocyte colony stimulating factor)
  G-CSF 300 units administered by trans-cervical infusion one time on day of human chorionic gonadotropin(hCG) trigger for Ovulation
- Saline Then G-CSF: Normal Saline
  Saline administered by trans-cervical infusion one time on day of hCG trigger for ovulation
Period: Cycle 1
Arm/Group | G-CSF Then Saline | Saline Then G-CSF
Started | 67 (Results reported In Barad et al 2014 are combined from both G-CSF studies) | 62 (Results reported In Barad et al 2014 are combined from both G-CSF studies)
Completed | 67 | 62
Not Completed | 0 | 0
Period: CrossoverCycle
Arm/Group | G-CSF Then Saline | Saline Then G-CSF
Started | 18 (16 ongoing pregnancies were not eligible for crossover, others chose to not have another IVF cycle) | 14 (14 ongoing pregnancies were not eligible for crossover, others chose to not have another IVF cycle)
Completed | 18 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- G-CSF Then Saline: G-CSF (Granulocyte colony stimulating factor)
  G-CSF 300 units administered by trans-cervical infusion one time on day of hCG trigger for Ovulation
  then
  Normal Saline
  Saline administered by trans-cervical infusion one time on day of hCG trigger for ovulation
- Saline Then G-CSF: Normal Saline
  Saline administered by trans-cervical infusion one time on day of hCG trigger for ovulation
  then
  G-CSF (Granulocyte colony stimulating factor)
  G-CSF 300 units administered by trans-cervical infusion one time on day of hCG trigger for Ovulation
- Total: Total of all reporting groups
Arm/Group | G-CSF Then Saline | Saline Then G-CSF | Total
Number analyzed (Participants) | 67 | 62 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 62 | 129
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 62 | 129
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 12 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 8 | 20
  White | 44 | 42 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 66 | 61 | 127
  Germany | 0 | 1 | 1
  United Kingdom | 1 | 0 | 1
AntiMulerian Hormone (AMH) [Mean (Standard Deviation); unit: ng/mL] | 2.07 (2.17) | 1.99 (2.38) | 2.03 (2.26)

OUTCOME MEASURES:

1. Primary Outcome: Embryo Implantation and Clinical Pregnancy Rates
Description: Implantation rate: The number of gestational sacs noted in the endometrial cavity 26 to 30 days after embryo transfer divided by the number of embryos transferred
  Clinical pregnancy:
  Gestational sac with evidence of a viable pregnancy at least 28 days after embryo transfer
Time Frame: 26 to 30 days after embryo transfer
Population: Presuming an implantation rate of 10% and anticipating a 10% increase to 20% with treatment, about 200 embryos transferred in each study arm would be needed for 80% power and alpha of 0.05.
Measure: Number; unit: Gestational sacs
Units Other Than Participants: Embryos Transferred
Groups:
- G-CSF: G-CSF (Granulocyte colony stimulating factor)
  G-CSF 300 units administered by trans-cervical infusion one time on day of hCG trigger for Ovulation
- Saline: Normal Saline
  Saline administered by trans-cervical infusion one time on day of hCG trigger for ovulation
Arm/Group | G-CSF | Saline
Number analyzed (Participants) | 81 | 80
Number analyzed (Embryos Transferred) | 212 | 207
Gestational sacs | 32 | 33
Statistical Analysis 1: Comparison: G-CSF vs Saline; Test type: Superiority or Other; p = 0.72, Cochran-Mantel-Haenszel

2. Secondary Outcome: Live Birth Rates
Description: Live birth rates among normal infertile couples undergoing IVF
Time Frame: Within nine months of embryo transfer
Measure: Number; unit: Live Birth
Arm/Group | G-CSF | Saline
Number analyzed (Participants) | 81 | 80
Live Birth | 22 | 19

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | G-CSF | Saline
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/80
Other Adverse Events (participants affected / at risk) | 0/81 | 0/80

LIMITATIONS AND CAVEATS:
The study results are applicable only to women undergoing routine IVF. Most of the women in this trial had normal endometrial thickness at randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No